CLINICAL TRIAL: NCT01962792
Title: A Multicenter Phase 1/2b Study of the Bruton's Tyrosine Kinase Inhibitor, Ibrutinib (PCI-32765), in Combination With Carfilzomib (Kyprolis™) in Subjects With Relapsed or Relapsed and Refractory Multiple Myeloma
Brief Title: Study of BTK Inhibitor, Ibrutinib in Combination With Carfilzomib in Subjects With Relapsed and Refractory Multiple Myeloma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Pharmacyclics LLC. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PCYC-1119-CA; Ibrutinib (PCI-32765)
Record Dates: First submitted 2013-09-27; First posted 2013-10-14 (Estimated); Results first posted 2021-12-21 (Actual); Last update posted 2021-12-21 (Actual); Status verified 2021-11

CONDITIONS: Multiple Myeloma
Keywords: PCI-32765; Multiple Myeloma; Relapsed Refractory Multiple Myeloma; Bruton's Tyrosine Kinase; Carfilzomib; Dexamethasone; Ibrutinib
MeSH Terms: conditions — Multiple Myeloma | interventions — ibrutinib; carfilzomib; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Phase 1 - Dose Finding (Experimental): Ibrutinib PO 560mg + Carfilzomib IV 20/27mg/m2 + Dexamethasone PO 20mg
  Interventions: Drug: Ibrutinib; Drug: Carfilzomib; Drug: Dexamethasone
- Phase 2b - Main Study (Experimental): Ibrutinib PO 560mg + Carfilzomib IV 20/36mg/m2 + Dexamethasone PO 20mg
  Interventions: Drug: Ibrutinib; Drug: Carfilzomib; Drug: Dexamethasone
- Phase 2b - Sub-study (Experimental): Ibrutinib PO 840 mg + Carfilzomib IV 20/36 mg/m2 + Dexamethasone PO 20 mg
  Interventions: Drug: Ibrutinib; Drug: Carfilzomib; Drug: Dexamethasone

INTERVENTIONS:
Drug: Ibrutinib
Drug: Carfilzomib
Drug: Dexamethasone

SUMMARY:
A MULTICENTER PHASE 1/2B STUDY OF THE BRUTON'S TYROSINE KINASE INHIBITOR, IBRUTINIB (PCI-32765), IN COMBINATION WITH CARFILZOMIB (KYPROLIS™) IN SUBJECTS WITH RELAPSED OR RELAPSED AND REFRACTORY MULTIPLE MYELOMA

DETAILED DESCRIPTION:
Bruton's tyrosine kinase (Btk) is an enzyme that is present in hematopoietic cells other than T cells and is necessary for downstream signal transduction from various hematopoietic receptors including the B cell receptor as well as some Fc, chemokine, and adhesion receptors, and is crucial for both B cell development and osteoclastogenesis. Although down-regulated in normal plasma cells, Btk is highly expressed in the malignant cells from many myeloma patients and some cell lines. PCI-32765 is a potent and specific inhibitor of Btk currently in Phase 2 and 3 clinical trials. The current study is designed and intended to determine the safety and efficacy of PCI-32765 in combination with carfilzomib (Kyprolis™) with and without dexamethasone in subjects with relapsed or relapsed and refractory multiple myeloma (MM).

ELIGIBILITY:
Inclusion Criteria:

* Measurable disease of MM as defined by at least ONE of the following:

  1. Serum monoclonal protein (SPEP) ≥1 g/dL
  2. Urine M-protein ≥200 mg/24 hrs
  3. Serum free light chain (SFLC): involved FLC ≥10 mg/dL (≥100 mg/L) AND abnormal kappa to lambda serum free light chain ratio
* Relapsed or relapsed and refractory MM after receiving at least 2 previous therapies, including an immunomodulator and bortezomib and had either no response or documented disease progression (according to IMWG criteria) to the most recent treatment regimen
* Adequate hematologic, hepatic, and renal function
* ECOG performance status of 0-2

Inclusion Criteria for Phase 2 Sub-study Cohort:

* Must meet all inclusion criteria defined in main study and in addition the following criteria must be met:
* Subject must have received a regimen containing carfilzomib in combination with dexamethasone as their most recent line of therapy and have:

  1. Achieved less than a partial response (<PR) following at least 4 cycles and are without evidence of progression disease (PD).

     OR
  2. Disease progression following an initial confirmed response of MR or better to the combination (according to IMWG response criteria).

Exclusion Criteria:

* Subject must not have primary refractory disease
* Plasma cell leukemia, primary amyloidosis or POEMS syndrome
* Unable to swallow capsules or disease significantly affecting gastrointestinal function
* Requires anti-coagulation with warfarin or a vitamin K antagonist
* Requires treatment with strong CYP3A inhibitors

Exclusion Criteria for Phase 2 Sub-study Cohort:

* Must not meet any exclusion criteria defined in main study except for exclusion criteria "Subject must not have primary refractory disease" which is related to prior carfilzomib

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2019-03 (Actual); Study Completion 2019-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (17):
- United States (16):
  - City of Hope, Duarte, California
  - University of California Los Angeles, Los Angeles, California
  - Colorado Blood Cancer Institute, Denver, Colorado
  - University of Nebraska Medical Center, Omaha, Nebraska
  - New York Presbyterian Hospital - Weill-Cornell, New York, New York
  - Mount Sinai Hospital, New York, New York
  - Carolinas Healthcare System, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - MUSC Hollings Cancer Center, Charleston, South Carolina
  - Vanderbilt Ingram Cancer Center, Nashville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Methodist Healthcare System, San Antonio, Texas
  - Virginia Commonwealth University, Richmond, Virginia
- McGill University, Montreal, Quebec, Canada

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 84 participants were enrolled and received at least 1 dose of study treatment (All-treated population); of these participants, a total of 59 received treatment at the recommended Phase 2 dose of study drug (All RP2D population).
Groups:
- Cohort 1 (560 mg): Ibrutinib PO 560mg + Carfilzomib IV 20/27 mg/m2
  Ibrutinib
  Carfilzomib
- Cohort 2a (560 mg): Ibrutinib PO 560 mg + Carfilzomib IV 20/36 mg/m2
  Ibrutinib
  Carfilzomib
- Cohort 2b (560 mg): Ibrutinib PO 560 mg+ Carfilzomib IV 20/36 mg/m2 Dexamethasone PO 20 mg
  Ibrutinib
  Carfilzomib
  Dexamethasone
- All RP2D (840 mg): Ibrutinib PO 840 mg + Carfilzomib IV 20/36 mg/m2 + Dexamethasone PO 20 mg
  Ibrutinib
  Carfilzomib
  Dexamethasone
Period: Overall Study
Arm/Group | Cohort 1 (560 mg) | Cohort 2a (560 mg) | Cohort 2b (560 mg) | All RP2D (840 mg)
Started | 3 | 5 | 17 | 59
Completed | 3 | 5 | 17 | 59
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 (560 mg) | Cohort 2a (560 mg) | Cohort 2b (560 mg) | All RP2D (840 mg) | Total
Number analyzed (Participants) | 3 | 5 | 17 | 59 | 84
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 1 | 12 | 33 | 46
  >=65 years | 3 | 4 | 5 | 26 | 38
Age, Continuous [Median (Standard Deviation); unit: years] | 69.0 (1.53) | 72.0 (9.21) | 60.0 (10.29) | 63.0 (9.86) | 63.5 (9.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 11 | 28 | 41
  Male | 2 | 4 | 6 | 31 | 43
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 2 | 7 | 10
  Not Hispanic or Latino | 2 | 5 | 15 | 51 | 73
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 3 | 5 | 17 | 59 | 84

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: -To evaluate the overall response (ORR) of ibrutinib in combination with carfilzomib and dexamethasone.
Time Frame: up to 4 years
Population: Please note that the analysis only includes participants who achieved the best response of complete response or partial response from the All-treated population (per protocol).
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 1 (560 mg): Ibrutinib PO 560 mg + Carfilzomib IV 20/27 mg/m2
  Ibrutinib
  Carfilzomib
Arm/Group | Cohort 1 (560 mg) | Cohort 2a (560 mg) | Cohort 2b (560 mg) | All RP2D (840 mg)
Number analyzed (Participants) | 3 | 5 | 17 | 59
Participants | 2 | 2 | 12 | 42

2. Secondary Outcome: Duration of Response (DOR)
Description: The time interval between the date of initial documentation of a response (PR or better) and the date of first documented evidence of progressive disease, death, or date of censoring for the subjects who had not progressed/died. The censoring date was the last adequate tumor assessment date.
Time Frame: Up to 4 years
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1 (560 mg) | Cohort 2a (560 mg) | Cohort 2b (560 mg) | All RP2D (840 mg)
Number analyzed (Participants) | 3 | 5 | 17 | 59
Months | 7.1 [1.2 to 13.0] | 15.3 [5.4 to 15.3] | 9.2 [3.0 to 14.5] | 7.2 [2.7 to 16.6]

3. Secondary Outcome: Overall Survival
Description: Time from date of first dose of study treatment to the date of death from any cause
Time Frame: Up to 4 years
Population: Please note that the analysis only includes participants who achieved the best response of complete response or partial response from the All RP2D population (per protocol).
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | All RP2D (840 mg)
Number analyzed (Participants) | 59
Months | 35.9 [0.9 to 51.8]

4. Secondary Outcome: Progression Free Survival (PFS)
Description: Time from date of first dose of study treatment to the date of first documented evidence of progressive disease, death or date of censoring for the subjects not progressed/died. The censoring date was the last adequate tumor assessment date.
Time Frame: Up to 4 years
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | All RP2D (840 mg)
Number analyzed (Participants) | 59
Months | 7.4 [4.6 to 10.2]

ADVERSE EVENTS:
Time Frame: 4 years, 2months
Description: The Deaths reported are Death during treatment and within 30 Days of Last Study Treatment.
Arm/Group | Cohort 1 (560 mg) | Cohort 2a (560 mg) | Cohort 2b (560 mg) | All RP2D (840 mg)
All-Cause Mortality (participants affected / at risk) | 0/3 | 4/5 | 9/17 | 22/59
Serious Adverse Events (participants affected / at risk) | 2/3 | 5/5 | 17/17 | 59/59
Other Adverse Events (participants affected / at risk) | 3/3 | 5/5 | 17/17 | 58/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (560 mg) (N=3) | Cohort 2a (560 mg) (N=5) | Cohort 2b (560 mg) (N=17) | All RP2D (840 mg) (N=59)
Pneumonia (Infections and infestations) | 1 (1) | 2 (2) | 1 | 6 (6)
Atrial Flutter (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 2
Left ventricular dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mitral valve disease (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Incarcerated umbilical hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 3 (3) | 2 (2)
Asthenia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Bronchopulmonary aspergillosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Escherichia bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Escherichia sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Necrotising Fasciitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pseudomonal sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tumor Lysis Syndrome (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Metastases to nervous sytem (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Non - small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headche (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pseudomonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastric haemmorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Acute haemorrhagic conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthritis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infection colitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia influenzal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pseudomonal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Staphylococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Viral Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Transfusion-related acute lung injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Deep Vein Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (560 mg) (N=3) | Cohort 2a (560 mg) (N=5) | Cohort 2b (560 mg) (N=17) | All RP2D (840 mg) (N=59)
Anaemia (Blood and lymphatic system disorders) | 1 | 3 | 6 | 24
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1 | 3 | 30
Atrial fibrillation (Cardiac disorders) | 1 | 1 | 2 | 2
Atrial flutter (Cardiac disorders) | 1 | 0 | 0 | 2
Constipation (Gastrointestinal disorders) | 1 | 2 | 5 | 14
Pyrexia (General disorders) | 1 | 3 | 8 | 12
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0 | 2 | 4
Influenza (Infections and infestations) | 1 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 7 | 17
Blood bilirubin increased (Investigations) | 1 | 0 | 0 | 6
Headache (Nervous system disorders) | 1 | 2 | 8 | 13
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 2 | 4
cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 7 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 2 | 6 | 16
Hypotension (Vascular disorders) | 1 | 0 | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 2 | 5
Left ventricular dysfunction (Cardiac disorders) | 0 | 1 | 1 | 1
Sinus bradycardia (Cardiac disorders) | 0 | 1 | 1 | 0
Eye swelling (Eye disorders) | 0 | 1 | 0 | 3
Diarrhoea (Gastrointestinal disorders) | 0 | 3 | 11 | 29
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 3 | 5
Flatulence (Gastrointestinal disorders) | 0 | 1 | 2 | 3
Vomiting (Gastrointestinal disorders) | 0 | 1 | 4 | 10
Chills (General disorders) | 0 | 3 | 1 | 7
Fatigue (General disorders) | 0 | 4 | 12 | 27
Malaise (General disorders) | 0 | 0 | 2 | 2
Asthenia (General disorders) | 0 | 1 | 1 | 3
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 4
Oedema peripheral (General disorders) | 0 | 1 | 0 | 17
Pain (General disorders) | 0 | 1 | 0 | 2
Drug hypersensitivity (Immune system disorders) | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 1 | 5
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 1 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 2
Skin infection (Infections and infestations) | 0 | 1 | 0 | 3
Urinary tract infection (Infections and infestations) | 0 | 1 | 5 | 8
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 2
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 5
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 6
Blood testosterone decreased (Investigations) | 0 | 1 | 0 | 0
Ejection fraction decreased (Investigations) | 0 | 1 | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 2 | 7 | 11
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 4 | 10
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0 | 10
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 16
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 3 | 3 | 13
Balance disorder (Nervous system disorders) | 0 | 1 | 2 | 1
Dizziness (Nervous system disorders) | 0 | 1 | 1 | 16
Memory impairment (Nervous system disorders) | 0 | 1 | 0 | 1
Tremor (Nervous system disorders) | 0 | 1 | 1 | 1
Confusional state (Psychiatric disorders) | 0 | 1 | 2 | 5
Haematuria (Renal and urinary disorders) | 0 | 1 | 1 | 2
Renal impairment (Renal and urinary disorders) | 0 | 1 | 1 | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 5 | 10
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 21
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 6 | 15
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 3 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 5
Increased tendency to bruise (Blood and lymphatic system disorders) | 0 | 0 | 2 | 7
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 1 | 2
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 4 | 3
Palpitations (Cardiac disorders) | 0 | 0 | 3 | 6
Mitral valve incompetence (Cardiac disorders) | 0 | 0 | 2 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 2 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 1 | 2
Aortic valve incompetence (Cardiac disorders) | 0 | 0 | 1 | 0
Atrial tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Left atrial dilatation (Cardiac disorders) | 0 | 0 | 1 | 0
Right atrial dilatation (Cardiac disorders) | 0 | 0 | 1 | 0
Supraventricular extrasystoles (Cardiac disorders) | 0 | 0 | 1 | 0
Tricuspid valve incompetence (Cardiac disorders) | 0 | 0 | 1 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 1 | 1
Middle ear effusion (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 1 | 0
Vision blurred (Eye disorders) | 0 | 0 | 2 | 4
Dry eye (Eye disorders) | 0 | 0 | 1 | 2
Lacrimation increased (Eye disorders) | 0 | 0 | 1 | 1
Ocular hyperaemia (Eye disorders) | 0 | 0 | 1 | 1
Periorbital oedema (Eye disorders) | 0 | 0 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 2 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 3 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 3 | 7
Nausea (Gastrointestinal disorders) | 0 | 0 | 8 | 26
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 3
Dental discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Diverticulum (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1 | 2
Eructation (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 13
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Melaena (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Oral disorder (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Oral dysaesthesia (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Oral pain (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Oral pruritus (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Palatal ulcer (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Pancreatic pseudocyst (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 8
Oedema peripheral (General disorders) | 0 | 0 | 4 | 0
Chest pain (General disorders) | 0 | 0 | 2 | 3
Gait disturbance (General disorders) | 0 | 0 | 2 | 3
Catheter site oedema (General disorders) | 0 | 0 | 1 | 0
Catheter site rash (General disorders) | 0 | 0 | 1 | 0
Oedema (General disorders) | 0 | 0 | 1 | 0
Feeling abnormal (General disorders) | 0 | 0 | 1 | 0
Localised oedema (General disorders) | 0 | 0 | 1 | 2
Systemic inflammatory response syndrome (General disorders) | 0 | 0 | 1 | 0
Peripheral swelling (General disorders) | 0 | 0 | 1 | 3
Hypersensitivity (Immune system disorders) | 0 | 0 | 1 | 0
Candida infection (Infections and infestations) | 0 | 0 | 1 | 2
Enterocolitis infectious (Infections and infestations) | 0 | 0 | 1 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 1 | 4
Catheter site infection (Infections and infestations) | 0 | 0 | 1 | 0
Fungal infection (Infections and infestations) | 0 | 0 | 1 | 1
Laryngitis (Infections and infestations) | 0 | 0 | 1 | 0
Onychomycosis (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia Fungal (Infections and infestations) | 0 | 0 | 1 | 0
Rash Pustular (Infections and infestations) | 0 | 0 | 1 | 0
Skin infection (Infections and infestations) | 0 | 0 | 1 | 0
Tinea pedis (Infections and infestations) | 0 | 0 | 1 | 0
Urinary tract infection bacterial (Infections and infestations) | 0 | 0 | 1 | 0
Vaginal infection (Infections and infestations) | 0 | 0 | 1 | 0
Animal bite (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Eyelid contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Post procedural contusion (Infections and infestations) | 0 | 0 | 1 | 1
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 2 | 4
Neutrophil count decreased (Investigations) | 0 | 0 | 2 | 2
Platelet count decreased (Investigations) | 0 | 0 | 2 | 7
White blood cell count decreased (Investigations) | 0 | 0 | 2 | 3
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 5
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 1 | 0
Brain natriuretic peptide increased (Investigations) | 0 | 0 | 1 | 0
Troponin increased (Investigations) | 0 | 0 | 1 | 0
Weight decreased (Investigations) | 0 | 0 | 1 | 2
Weight increased (Investigations) | 0 | 0 | 1 | 0
Hypocalcaemia (Investigations) | 0 | 0 | 4 | 0
Dehydration (Infections and infestations) | 0 | 0 | 3 | 3
Hyperglycaemia (Investigations) | 0 | 0 | 3 | 10
Hypomagnesaemia (Investigations) | 0 | 0 | 2 | 3
Electrolyte imbalance (Investigations) | 0 | 0 | 1 | 0
Diabetes mellitus (Investigations) | 0 | 0 | 1 | 0
Fluid overload (Investigations) | 0 | 0 | 1 | 0
Hyperkalaemia (Investigations) | 0 | 0 | 1 | 4
Hypertriglyceridaemia (Investigations) | 0 | 0 | 1 | 0
Hyperuricaemia (Investigations) | 0 | 0 | 1 | 6
Hypoalbuminaemia (Investigations) | 0 | 0 | 1 | 6
Hyponatraemia (Investigations) | 0 | 0 | 1 | 9
Hypophosphataemia (Investigations) | 0 | 0 | 1 | 5
Lactic acidosis (Investigations) | 0 | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 5 | 5
Arthralgia (Investigations) | 0 | 0 | 4 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 4 | 9
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 8
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 2
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 3
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Soft tissue mass (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 3 | 4
Dysgeusia (Nervous system disorders) | 0 | 0 | 3 | 3
Depressed level of consciousness (Nervous system disorders) | 0 | 0 | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 1 | 2
Insomnia (Psychiatric disorders) | 0 | 0 | 5 | 18
Anxiety (Psychiatric disorders) | 0 | 0 | 3 | 3
Depression (Psychiatric disorders) | 0 | 0 | 2 | 3
Hallucination (Psychiatric disorders) | 0 | 0 | 2 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 1 | 1
Disorientation (Psychiatric disorders) | 0 | 0 | 1 | 0
Irritability (Psychiatric disorders) | 0 | 0 | 1 | 1
Mania (Psychiatric disorders) | 0 | 0 | 1 | 0
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 1 | 3
Chronic kidney disease (Renal and urinary disorders) | 0 | 0 (0) | 2 | 0
Incontinence (Renal and urinary disorders) | 0 | 0 | 1 | 1
Urinary retention (Renal and urinary disorders) | 0 | 0 | 1 | 1
Genital rash (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Rales (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 4 | 4
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 6
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 3
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 3
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 3
Lower respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 4 | 1
Rash maculo-papular (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 4 | 4
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 3 | 3
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 3 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 3
Skin fissures (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 4
Nail ridging (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Flushing (Vascular disorders) | 0 | 0 | 2 | 2
Hot flush (Vascular disorders) | 0 | 0 | 2 | 1
Aortic dilatation (Vascular disorders) | 0 | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 1
Venous thrombosis (Vascular disorders) | 0 | 0 | 1 | 1
Phlebitis (Vascular disorders) | 0 | 0 | 0 | 2
Jugular vein distension (Vascular disorders) | 0 | 0 | 0 | 1
Thrombophlebitis (Vascular disorders) | 0 | 0 | 0 | 1
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Skin mass (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Scab (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Hair disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 3
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Uterine prolapse (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Testicular cyst (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Scrotal oedema (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Vulvovaginal discomfort (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Urinary hesitation (Renal and urinary disorders) | 0 | 0 | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 4
Mood swings (Psychiatric disorders) | 0 | 0 | 0 | 1
Mood altered (Psychiatric disorders) | 0 | 0 | 0 | 1
Anxiety disorder (Psychiatric disorders) | 0 | 0 | 0 | 1
Psychotic disorder (Psychiatric disorders) | 0 | 0 | 0 | 2
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 1
Peroneal nerve palsy (Nervous system disorders) | 0 | 0 | 0 | 1
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 1
Migraine (Nervous system disorders) | 0 | 0 | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 1
Ataxia (Nervous system disorders) | 0 | 0 | 0 | 1
Aphonia (Nervous system disorders) | 0 | 0 | 0 | 1
Amnesia (Nervous system disorders) | 0 | 0 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 2
Coordination abnormal (Nervous system disorders) | 0 | 0 | 0 | 2
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 4
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 11
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2
Joint lock (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 9
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hyperammonaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Fluid retention (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Enzyme abnormality (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2
Hypocalcaemia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 5
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 5
White blood cell count increased (Investigations) | 0 | 0 | 0 | 1
Transaminases increased (Investigations) | 0 | 0 | 0 | 1
Platelet count increased (Investigations) | 0 | 0 | 0 | 1
Lipase increased (Investigations) | 0 | 0 | 0 | 1
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 1
Electrocardiogram ST-T segment depression (Investigations) | 0 | 0 | 0 | 1
Blood uric acid decreased (Investigations) | 0 | 0 | 0 | 1
Blood phosphorus increased (Investigations) | 0 | 0 | 0 | 1
Bilirubin conjugated increased (Investigations) | 0 | 0 | 0 | 1
Urine output decreased (Investigations) | 0 | 0 | 0 | 2
Cardiac murmur (Investigations) | 0 | 0 | 0 | 2
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 3
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 4
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 4
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 5
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Tooth infection (Infections and infestations) | 0 | 0 | 0 | 1
Staphylococcal skin infection (Infections and infestations) | 0 | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 1
Oral infection (Infections and infestations) | 0 | 0 | 0 | 1
Oral bacterial infection (Infections and infestations) | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 1
Nail infection (Infections and infestations) | 0 | 0 | 0 | 1
Mucosal infection (Infections and infestations) | 0 | 0 | 0 | 1
Lymph gland infection (Infections and infestations) | 0 | 0 | 0 | 1
Localised infection (Infections and infestations) | 0 | 0 | 0 | 1
Infusion site cellulitis (Infections and infestations) | 0 | 0 | 0 | 1
Herpes simplex (Infections and infestations) | 0 | 0 | 0 | 1
Furuncle (Infections and infestations) | 0 | 0 | 0 | 1
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 1
Endocarditis bacterial (Infections and infestations) | 0 | 0 | 0 | 1
Ecthyma (Infections and infestations) | 0 | 0 | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 1
Device related infection (Infections and infestations) | 0 | 0 | 0 | 1
Cytomegalovirus infection (Infections and infestations) | 0 | 0 | 0 | 1
Cystitis (Infections and infestations) | 0 | 0 | 0 | 1
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 0 | 1
Catheter site pustule (Infections and infestations) | 0 | 0 | 0 | 1
Bronchitis viral (Infections and infestations) | 0 | 0 | 0 | 1
Acute sinusitis (Infections and infestations) | 0 | 0 | 0 | 1
Acute haemorrhagic conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 1
Rhinovirus infection (Infections and infestations) | 0 | 0 | 0 | 2
Respiratory syncytial virus infection (Infections and infestations) | 0 | 0 | 0 | 2
Ear infection (Infections and infestations) | 0 | 0 | 0 | 2
Corona virus infection (Infections and infestations) | 0 | 0 | 0 | 2
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 2
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 3
Rash pustular (Infections and infestations) | 0 | 0 | 0 | 3
Hypogammaglobulinaemia (Immune system disorders) | 0 | 0 | 0 | 2
Hepatomegaly (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 0 | 5
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 1
Infusion site reaction (General disorders) | 0 | 0 | 0 | 1
Feeling jittery (General disorders) | 0 | 0 | 0 | 1
Facial pain (General disorders) | 0 | 0 | 0 | 1
Catheter site pain (General disorders) | 0 | 0 | 0 | 1
Catheter site erythema (General disorders) | 0 | 0 | 0 | 1
Injection site bruising (General disorders) | 0 | 0 | 0 | 2
Face oedema (General disorders) | 0 | 0 | 0 | 2
Chest discomfort (General disorders) | 0 | 0 | 0 | 2
Influenza like illness (General disorders) | 0 | 0 | 0 | 7
Salivary hypersecretion (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Oesophageal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Hypoaesthesia oral (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Anal incontinence (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Presbyopia (Eye disorders) | 0 | 0 | 0 | 1
Eye pruritus (Eye disorders) | 0 | 0 | 0 | 1
Eye pain (Eye disorders) | 0 | 0 | 0 | 1
Eye irritation (Eye disorders) | 0 | 0 | 0 | 1
Eye haemorrhage (Eye disorders) | 0 | 0 | 0 | 1
Diplopia (Eye disorders) | 0 | 0 | 0 | 1
Blepharospasm (Eye disorders) | 0 | 0 | 0 | 1
Visual impairment (Eye disorders) | 0 | 0 | 0 | 2
Hypoparathyroidism (Endocrine disorders) | 0 | 0 | 0 | 1
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 0 | 1
Cushingoid (Endocrine disorders) | 0 | 0 | 0 | 2
Tympanic membrane perforation (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Middle ear inflammation (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Cerumen impaction (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 2
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Cardiac flutter (Cardiac disorders) | 0 | 0 | 0 | 1
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 4
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 7
Conjunctivitis Viral (Infections and infestations) | 0 | 0 | 0 | 1
Eye Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Urinary Incontinence (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastroenteritis Viral (Infections and infestations) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-09-05): https://cdn.clinicaltrials.gov/large-docs/92/NCT01962792/Prot_SAP_000.pdf